CLINICAL TRIAL: NCT03304158
Title: Community Based Intervention for Management of Diabetes in Nepal (COBIN-D): A Cluster Randomised Controlled Trial
Brief Title: Community Based Management of Diabetes in Nepal
Acronym: COBIN-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Bishal Gyawali, PhD scholar, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AUBIS123
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Non-communicable disease; Primary health care; Nepal
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCHV visit-diabetes (Experimental)
  Interventions: Behavioral: FCHV visit
- FCHV no visit-diabetes (No Intervention)

INTERVENTIONS:
Behavioral: FCHV visit — FCHVs will visit selected households 3 times a year for providing health promotion messages and measure the blood glucose
  Arms: FCHV visit-diabetes

SUMMARY:
Type 2 diabetes is the largest growing concern across the globe, and this is particularly apparent in developing countries, including Nepal. Despite the growing burden and chronic nature of diabetes, prevention and control of this disease is far from adequate setting in Nepal. Moreover, there is lack of evidence on effectiveness and affordability of a population approach on reducing blood glucose level among diabetes persons. The main aim of this study is to determine the effect of Female Community Health Volunteers' (FCHVs)-led family-based health education and screening on blood sugar level in adults at community level in Nepal. This is a community-based cluster randomized controlled trial involving family based health education through FCHVs in Nepal. People ≥25 years of age listed in the Community-Based Management of Hypertension (COBIN) study and who were diabetics are eligible for eligible for participation in the study. FCHVs will conduct family based health education and fasting blood glucose measurements in the treatment arm vs not any interventions in the control arm. Independent assessors will conduct the baseline and end line assessment of the intervention. Intention to treat analysis and per protocol analysis will be used in analysis to detect significant differences between treatment and control group participants at baseline and follow up. For individual outcomes, proportions will be compared using Chi-square test and continuous measures will be compared using t-tests. Random effect mixed regression analysis will be adjusted for age and sex. Since randomisation will be at the cluster level in the study, a random-effect model will be used to account for clustering effect. Effectiveness of the intervention will be tested by analysis of covariance, which will allow us to adjust for baseline differences between groups. It is anticipated that the study can give valuable information regarding effectiveness, acceptability, and feasibility of an innovative way to improve diabetes management. Assessing the FCHVs' ability to address diabetes may contribute to develop a policy that can be scaled-up to a national level.

ELIGIBILITY:
Inclusion Criteria:

* Those ≥25 years of age and listed in the COBIN study
* Those who participated in our prevalence study
* Those who give consent to participate in our intervention study
* Those who do not have any plan to migrate from the study area for at least 1 year
* Those who are non-pregnant women
* Those who are not severely ill

Exclusion Criteria:

* Those who do not give consent
* Those who are pregnant women
* Those who are severely ill
* Those who have plans to migrate from the study area within 1 year

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Mean fasting blood glucose level | 1 year
  Change in mean fasting blood glucose level in diabetes populations

CONTACTS AND LOCATIONS:
Locations (1):
- A semi-urban area of Pokhara-Lekhnath Metropolitan City of Nepal, Pokhara, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyawali B, Sharma R, Mishra SR, Neupane D, Vaidya A, Sandbaek A, Kallestrup P. Effectiveness of a Female Community Health Volunteer-Delivered Intervention in Reducing Blood Glucose Among Adults With Type 2 Diabetes: An Open-Label, Cluster Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2035799. doi: 10.1001/jamanetworkopen.2020.35799. PMID 33523189
- [Derived] Gyawali B, Neupane D, Vaidya A, Sandbaek A, Kallestrup P. Community-based intervention for management of diabetes in Nepal (COBIN-D trial): study protocol for a cluster-randomized controlled trial. Trials. 2018 Oct 22;19(1):579. doi: 10.1186/s13063-018-2954-3. PMID 30348188